CLINICAL TRIAL: NCT01147588
Title: An Open-label, Randomized, 4-treatment, 3-period, Crossover Interaction Study, Evaluating the Effect of Esomeprazole 40 mg, Omeprazole 80 mg or Lansoprazole 60 mg on the Pharmacodynamics and the Pharmacokinetics of Clopidogrel in Healthy Volunteers
Brief Title: Study Evaluating Effect of Esomeprazole, Omeprazole or Lansoprazole on the Pharmacodynamics (PD) and Pharmacokinetics (PK) of Clopidogrel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D9612C00034
Record Dates: First submitted 2010-06-04; First posted 2010-06-22 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Healthy
Keywords: open label; randomized; 4-treatment; 3-period; crossover; interaction study; Safety; tolerability; pharmacokinetics; pharmacodynamics
MeSH Terms: interventions — Lansoprazole; Omeprazole; Esomeprazole; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): lansoprazole 60 mg + clopidogrel 300 mg/ 75 mg
  Interventions: Drug: lansoprazole; Drug: clopidogrel
- 2 (Experimental): omeprazole 80 mg + clopidogrel 300/75 mg
  Interventions: Drug: omeprazole; Drug: clopidogrel
- 3 (Experimental): esomeprazole 40 mg + clopidogrel 300/75 mg
  Interventions: Drug: esomeprazole; Drug: clopidogrel
- 4 (Experimental): clopidogrel 300/75 mg alone
  Interventions: Drug: clopidogrel

INTERVENTIONS:
Drug: lansoprazole — 60 mg (2x30-mg capsule), once daily
  Arms: 1
Drug: omeprazole — 80 mg (2x40-mg capsule), once daily
  Arms: 2
Drug: esomeprazole — 40 mg (1x40-mg capsule), once daily
  Arms: 3
Drug: clopidogrel — 300 mg loading dose on Day 1 then 75 mg daily for 28 days

SUMMARY:
The aim of this study is to determine if there is a pharmacological interaction between clopidogrel and different types of proton pump inhibitors (PPIs), and if the extent of this possible interaction would change over time.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males within the age of 18-45 years and females within the age of 18-55 years with suitable veins for cannulation or repeated vein puncture. Females must be of non-childbearing potential.
* Weight of 50-95kg, inclusive, and a BMI between 19-30 kg/m2, inclusive.
* No clinically significant abnormal findings as judged by the Investigator on enrollment physical exam.

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in study.
* History or presence of gastrointestinal e.g. GI ulcer, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs.
* Any clinically significant illness within 4 weeks of the first administration of investigational product. Any medical/surgical procedure or trauma within 3 months of the treatment period; scheduled surgery, including dental surgery within 2 weeks.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 149 (Actual)
Dates: Start 2010-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Assess the effect of esomeprazole 40 mg, omeprazole 80 mg or lansoprazole 60 mg on the PK profile of clopidogrel active metabolite by assessing the inhibition of platelet aggregation (mIPA). | Baseline
Assess the effect of esomeprazole 40 mg, omeprazole 80 mg or lansoprazole 60 mg on the PK profile of clopidogrel active metabolite by assessing the inhibition of platelet aggregation (mIPA). | Day 2
Assess the effect of esomeprazole 40 mg, omeprazole 80 mg or lansoprazole 60 mg on the PK profile of clopidogrel active metabolite by assessing the inhibition of platelet aggregation (mIPA). | Day 6
Assess the effect of esomeprazole 40 mg, omeprazole 80 mg or lansoprazole 60 mg on the PK profile of clopidogrel active metabolite by assessing the inhibition of platelet aggregation (mIPA). | Day 15
Assess the effect of esomeprazole 40 mg, omeprazole 80 mg or lansoprazole 60 mg on the PK profile of clopidogrel active metabolite by assessing the inhibition of platelet aggregation (mIPA). | Day 30

SECONDARY OUTCOMES:
Assess the effect of esomeprazole 40 mg, omeprazole 80 mg or lansoprazole 60 mg on the PK profile of clopidogrel active metabolite by assessing the AUC, AUC 0-t and Cmax after the loading dose of clopidogrel (Day 1) and AUC 0-t, ss and Css, max. | Days 5,14, 29
Evaluate the safety and tolerability of clopidogrel given concomittantly with esomeprazole, omeprazole or lansoprazole by assessment of adverse events and calculation of change from baseline for clinical laboratory tests, vital signs and pECG. | Every in-house day

CONTACTS AND LOCATIONS:
Overall Officials: Kelli Craven, MD, Principal Investigator — Quintiles, Inc.; Ken Price, Study Director — AstraZeneca; Mirjana Kujacic, Study Chair — AstraZeneca
Locations (1):
- Research Site, Overland Park, Kansas, United States

REFERENCES:
- [Derived] Andersson T, Nagy P, Niazi M, Nylander S, Galbraith H, Ranjan S, Wallentin L. Effect of esomeprazole with/without acetylsalicylic acid, omeprazole and lansoprazole on pharmacokinetics and pharmacodynamics of clopidogrel in healthy volunteers. Am J Cardiovasc Drugs. 2014 Jun;14(3):217-27. doi: 10.1007/s40256-014-0073-4. PMID 24677117